CLINICAL TRIAL: NCT04044300
Title: A Prospective, Randomized Controlled Trial Comparing Percutaneous Screw Fixation to Non-Operative Management for the Treatment of Sacral Fragility Fractures
Brief Title: Operative vs Non-Operative Treatment of Sacral Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: More Foundation (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3209
Record Dates: First submitted 2019-04-30; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Sacral Fracture
Keywords: sacral fracture, function, pain
MeSH Terms: conditions — Pain | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to one of two treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative (Experimental): A single trans-iliac, trans-sacral screw will be inserted at the sacral one or sacral two level.
  Interventions: Procedure: Single screw fixation
- Non-operative (Experimental): Continued pain management and physical therapy
  Interventions: Procedure: Single screw fixation; Other: Conservative

INTERVENTIONS:
Procedure: Single screw fixation — A single trans-iliac, trans-sacral screw will be inserted at the sacral one or sacral two level based upon fracture location.
Other: Conservative — Continued pain management and physical therapy.
  Arms: Non-operative

SUMMARY:
The purpose of this study is to compare percutaneous trans-iliac trans-sacral screw fixation to non-operative management for the treatment of symptomatic, sacral fragility fractures in elderly patients.

DETAILED DESCRIPTION:
Sacral fragility fractures cause significant pain and morbidity in the elderly population in which they occur. These low-energy pelvic injuries can cause prolonged immobility, long hospital stays, and requirement for higher levels of care.

Subjects will undergo a 48 hour period of physical therapy and pain management following identification of the sacral fracture.. If the subject has substantial pain or disability, the subject is eligible for enrollment in the RCT and randomization of 1:1 to one of two groups.

Group 1: Operative treatment: A single trans iliac trans sacral screw will be inserted at the sacral one or sacral two level based upon fracture location.

Group 2: Conservative (non-operative) treatment: Continued pain management and physical therapy advanced with weight bearing as tolerated.

The purpose of this study is to compare percutaneous trans-iliac trans-sacral screw fixation to non-operative management for the treatment of symptomatic, sacral fragility fractures in elderly patients.

Primary Objective: To compare the functional outcome and pain in elderly patients surgically treated compared to those non-operatively treated for sacral fractures.

Secondary Objective: To compare discharge disposition, length of stay in care facility post-discharge, complications, and need for ambulatory aid in elderly patients surgically treated compared to those non-operatively treated for sacral fractures.

Hypothesis: Subjects in the operative group will have improvement in functional outcome and pain at 2 weeks, higher likelihood of discharge to independent living, shorter stays in care facilities post-discharge, less complications, and less need for ambulatory aids.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 60 years of age
2. Pelvic ring fractures classified as LC1 or sacral U, confirmed with plain radiographs, CT and/or MRI
3. Fracture is the result of a low energy mechanism of injury or an insufficiency fracture without a precipitating event
4. Onset of symptoms within four weeks of presentation to hospital
5. Significant pain or disability determined by:

   1. Reported pain score ≥ 7 using the Visual Analogue Score (VAS) after a Timed "Up & Go" (TUG) test, or
   2. Inability to complete the TUG test
   3. Inability to get out of bed secondary to pain for 2 consecutive days

Exclusion Criteria:

1. Vertically or rotationally unstable pelvic ring injuries
2. Pathologic fracture secondary to tumor
3. Non-ambulatory prior to injury
4. Acute neurologic deficit
5. High-energy mechanism of injury
6. Concomitant lower extremity fractures affecting ambulation
7. Presence of another injury or medical condition that prevents ambulation
8. Presence of hardware or sacral morphology that prevents percutaneous sacral fixation
9. Enrollment in another research study that precludes co-enrollment
10. Inability to speak English
11. Dementia with inability to answer questions and participate in study
12. Likely problems, in the judgment of the investigators, with maintaining follow-up (i.e. patients with no fixed address, not mentally competent to give consent, intellectually challenged patients without adequate support, etc.)
13. Incarcerated or pending incarceration

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) Test | 2 weeks
  TUG Test
Sacral Region Pain | 2 weeks
  Visual Analog Pain Scale, minimum score 0, maximum score 10, from no pain to worst possible pain

SECONDARY OUTCOMES:
Discharge Disposition Location | Up to 21 days
  Location that subject was discharged to at hospital discharge: Home, Rehabilitation, Skilled Nursing Facility
Facility Length of Stay | Up to 21 days
  Number of days in a rehabilitation or skilled nursing facility after hospital discharge
Ambulatory aid | 2 weeks
  Use of walker, cane, or wheelchair
Complications | Up to 1 year
  Screw migration, secondary surgery related to primary procedure, neurological deficit related to screw insertion, surgical site infection, wound dehiscence, deep infection, related re-admission, decubitus ulcer, pneumonia, deep vein thrombosis, pulmonary embolism, death
Patient Reported Health Outcome | Change from baseline to 1 year
  Veterans Rand 12-item Health Survey (VR-12). This is a health related quality of life survey with 2 scores, Physical Component Score (PCS) including general health, physical functioning, physical role accomplishment, bodily pain and Mental Component Score (MCS) including role-emotional, vitality/mental health, social functioning. The results of the VR-12 are reported as 2 scores, MCS and PCS. The score range is 0-100 for each score, where a 0 score indicates the lowest level of health and a score of 100 indicates the highest level of health. The US population average PCS and MCS are both 50 points. The standard deviation is 10 points.
Patient Reported Outcome | Change from baseline to 1 year
  Hip dysfunction and Osteoarthritis Outcome Score (HOOS), Total score of 0-100 with higher scores representing better function

OTHER OUTCOMES:
Hospital length of stay | Up to 21 days
  Number of days hospitalized
Narcotic use | 2 weeks
  Use of narcotic pain medication, total in milligram equivalents
Healing | Change in healing from baseline to 1 year
  Standard pelvic radiographs (AP, inlet, outlet, and lateral sacral views) will be performed to evaluate radiographic outcomes such as fracture healing, fixation failure, and fracture displacement.

CONTACTS AND LOCATIONS:
Overall Officials: Clifford B Jones, MD, Principal Investigator — The CORE Institute
Locations (1):
- The CORE Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newhouse KE, el-Khoury GY, Buckwalter JA. Occult sacral fractures in osteopenic patients. J Bone Joint Surg Am. 1992 Dec;74(10):1472-7. PMID 1364816
- [Background] Wild A, Jaeger M, Haak H, Mehdian SH. Sacral insufficiency fracture, an unsuspected cause of low-back pain in elderly women. Arch Orthop Trauma Surg. 2002 Feb;122(1):58-60. doi: 10.1007/s004020100333. PMID 11995886
- [Background] Grasland A, Pouchot J, Mathieu A, Paycha F, Vinceneux P. Sacral insufficiency fractures: an easily overlooked cause of back pain in elderly women. Arch Intern Med. 1996 Mar 25;156(6):668-74. doi: 10.1001/archinte.156.6.668. PMID 8629880
- [Background] Galbraith JG, Butler JS, Blake SP, Kelleher G. Sacral insufficiency fractures: an easily overlooked cause of back pain in the ED. Am J Emerg Med. 2011 Mar;29(3):359.e5-6. doi: 10.1016/j.ajem.2010.04.015. Epub 2010 Aug 2. PMID 20675092
- [Background] Dasgupta B, Shah N, Brown H, Gordon TE, Tanqueray AB, Mellor JA. Sacral insufficiency fractures: an unsuspected cause of low back pain. Br J Rheumatol. 1998 Jul;37(7):789-93. doi: 10.1093/rheumatology/37.7.789. PMID 9714359
- [Background] Isdale AH. Sacral insufficiency fractures: an unsuspected cause of low back pain. Rheumatology (Oxford). 1999 Jan;38(1):90. doi: 10.1093/rheumatology/38.1.90a. No abstract available. PMID 10334691
- [Background] Lin JT, Lane JM. Sacral stress fractures. J Womens Health (Larchmt). 2003 Nov;12(9):879-88. doi: 10.1089/154099903770948104. PMID 14670167
- [Background] Lourie H. Spontaneous osteoporotic fracture of the sacrum. An unrecognized syndrome of the elderly. JAMA. 1982 Aug 13;248(6):715-7. PMID 7097924
- [Background] Mears SC, Berry DJ. Outcomes of displaced and nondisplaced pelvic and sacral fractures in elderly adults. J Am Geriatr Soc. 2011 Jul;59(7):1309-12. doi: 10.1111/j.1532-5415.2011.03455.x. Epub 2011 Jun 30. PMID 21718260
- [Background] Tsiridis E, Upadhyay N, Giannoudis PV. Sacral insufficiency fractures: current concepts of management. Osteoporos Int. 2006 Dec;17(12):1716-25. doi: 10.1007/s00198-006-0175-1. Epub 2006 Jul 20. PMID 16855863
- [Background] Rommens PM, Hofmann A. Comprehensive classification of fragility fractures of the pelvic ring: Recommendations for surgical treatment. Injury. 2013 Dec;44(12):1733-44. doi: 10.1016/j.injury.2013.06.023. Epub 2013 Jul 18. PMID 23871193
- [Background] Sanders D, Fox J, Starr A, Sathy A, Chao J. Transsacral-Transiliac Screw Stabilization: Effective for Recalcitrant Pain Due to Sacral Insufficiency Fracture. J Orthop Trauma. 2016 Sep;30(9):469-73. doi: 10.1097/BOT.0000000000000596. PMID 27551916
- [Background] Walker JB, Mitchell SM, Karr SD, Lowe JA, Jones CB. Percutaneous Transiliac-Transsacral Screw Fixation of Sacral Fragility Fractures Improves Pain, Ambulation, and Rate of Disposition to Home. J Orthop Trauma. 2018 Sep;32(9):452-456. doi: 10.1097/BOT.0000000000001243. PMID 29916895
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Sembler Soles GL, Lien J, Tornetta P 3rd. Nonoperative immediate weightbearing of minimally displaced lateral compression sacral fractures does not result in displacement. J Orthop Trauma. 2012 Oct;26(10):563-7. doi: 10.1097/BOT.0b013e318251217b. PMID 22495523
- [Background] Eckardt H, Egger A, Hasler RM, Zech CJ, Vach W, Suhm N, Morgenstern M, Saxer F. Good functional outcome in patients suffering fragility fractures of the pelvis treated with percutaneous screw stabilisation: Assessment of complications and factors influencing failure. Injury. 2017 Dec;48(12):2717-2723. doi: 10.1016/j.injury.2017.11.002. Epub 2017 Nov 4. PMID 29122281
- [Background] Kennedy DM, Stratford PW, Wessel J, Gollish JD, Penney D. Assessing stability and change of four performance measures: a longitudinal study evaluating outcome following total hip and knee arthroplasty. BMC Musculoskelet Disord. 2005 Jan 28;6:3. doi: 10.1186/1471-2474-6-3. PMID 15679884
- [Background] Gautschi OP, Stienen MN, Corniola MV, Joswig H, Schaller K, Hildebrandt G, Smoll NR. Assessment of the Minimum Clinically Important Difference in the Timed Up and Go Test After Surgery for Lumbar Degenerative Disc Disease. Neurosurgery. 2017 Mar 1;80(3):380-385. doi: 10.1227/NEU.0000000000001320. PMID 27352275